CLINICAL TRIAL: NCT05381831
Title: The Effects of Intranasal Testosterone (NatestoTM) for Treatment of Hypogonadism on Maintenance of Spermatogenesis
Brief Title: Natesto Spermatogenesis Reboot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202102979; OCR41644 (Other: UF OnCore)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NatestoTM (Experimental): Participants in this group will receive Natesto for a 26 consecutive weeks treatment course
  Interventions: Drug: NatestoTM

INTERVENTIONS:
Drug: NatestoTM — Administering daily intranasal testosterone, Natesto nasal gel is available as a metered-dose pump. One pump actuation delivers 5.5 mg of testosterone

SUMMARY:
This is a prospective, non-blinded study of hypogonadal men with a history of testosterone therapy who became azoospermic or severely oligospermic and wish to avoid symptoms of hypogonadism during their recovery of spermatogenesis in an effort to establish paternity. The study will determine if Natesto can alleviate hypogonadal symptoms while preserving the recovery of spermatogenesis

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 64 years of age, with documented onset of testosterone induced hypogonadism with impaired semen parameters who are attempting to achieve a successful pregnancy.
* Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
* Serum total testosterone < 350 ng/dL based on 2 consecutive blood samples obtained 1-4 weeks apart between 6 and 10 AM following an appropriate washout of current androgen replacement therapy; with clinical symptoms of hypogonadism such as diminished energy and sexual function; and/or a decreased sperm count (<20 million sperm/mL semen).
* Discontinued current testosterone replacement treatment and completed a washout of 4 weeks following androgen treatment (excluding Testopel TM). Washout must be completed prior to collection of baseline serum testosterone samples to determine study eligibility.
* Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, and laboratory profile.

Exclusion Criteria:

* History of significant sensitivity or allergy to androgens, castor oil or product excipients.
* Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up.
* Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or I-PSS score greater than 19 points.
* Body mass index (BMI) equal to or greater than or equal to 40 kg/m2.
* History of vasectomy.
* Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

  1. Baseline hemoglobin greater than 16 g/dL
  2. Hematocrit less than 35% or greater than 50%
  3. PSA greater than 4 ng/mL and age greater than 40
* History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
* History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.
* History of stroke or myocardial infarction within the past 5 years.
* History of, or current or suspected, prostate or breast cancer.
* History of diagnosed, severe, untreated, obstructive sleep apnea.
* History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
* History of nasal disorders such as nasal polyps; nasal septal perforation; nasal surgery; nasal trauma resulting in nasal fracture within the previous 6 months or nasal fracture that caused a deviated anterior nasal septum; sinus surgery or sinus disease
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 12 weeks prior to the start of treatment.
* Inadequate venous access for collection of serial blood samples required for pharmacokinetic profiles.
* Receipt of any investigational product within 4 weeks or within 5 half-lives prior to the start of treatment.
* Inability to understand and provide written informed consent for the study.
* Considered by the investigator or the sponsor-designated physician, for any reason, that the subject is an unsuitable candidate to receive Natesto.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The condition only affects males
Enrollment: 13 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Changes in total motile sperm count | Baseline up to 26 weeks
  Change in sperm count will be analyzed using the ANOVA. A change in < ± 10% will be reject the null hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Campbell, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT05381831/ICF_000.pdf